CLINICAL TRIAL: NCT00277979
Title: Utilization of 3D Echocardiography in the Management of Infantile Pompe's Disease: Two Case Reports
Brief Title: 3D Echocardiography Managing Infantile Pompe's Disease
Status: Terminated | Type: Observational
Why Stopped: project withdrawn
Sponsor: Children's Healthcare of Atlanta (Other)
Responsible Party: Chairman, Children's Healthcare of Atlanta Institutional Review Board
Other Study IDs: 05-058
Record Dates: First submitted 2006-01-13; First posted 2006-01-18 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2007-12

CONDITIONS: Congenital Disorders
Keywords: pediatric; cardiac; Infantile Pompe's Disease; 3D Echocardiography
MeSH Terms: conditions — Congenital, Hereditary, and Neonatal Diseases and Abnormalities

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Pompe's disease, also known as glycogen storage disease type II, is a genetic disorder due to deficiency of acid glucosidase (GAA), which results in lysosomal glycogen storage in various tissues.

Very low levels of GAA usually present in infancy, lead to a progressive cardiac and skeletal muscle disorder and death before age 1 year.

Most infants develop massive hypertrophic cardiomyopathy which progresses to dilated cardiomyopathy and cardiorespiratory arrest.

3D echocardiography can be a simple, non-invasive method of following cardiac disease progression in infantile Pompe's disease.

DETAILED DESCRIPTION:
We report the utilization of real-time 3D echocardiography and new in-line software to calculate cardiac mass, volume and function in two cases of infantile Pompe's Disease. Furthermore, the multi-dimension cine loop showed the severity of cavity obliteration during the cardiac cycle.

We present 2 cases seen at our institution between January - February, 2005 in infants ages 1 and 5 months, both with cardiac signs as initial presentation. The younger infant had cardiomegaly since birth and was hospitalized briefly for respiratory distress at 1 month. The older infant, diagnosed at 4 months with hypertrophic cardiomyopathy, was hospitalized after cardiac arrest one month later. Both children had various tests done during the course of diagnosis and treatment, including GAA enzyme assay, cardiac catheterization, endomyocardial biopsy, developmental assessment, genetic evaluation, EKG, CXR and echocardiography.

ELIGIBILITY:
Inclusion Criteria:

* Infant seen at Children's Healthcare of Atlanta, Egleston January - February, 2005 Infantile Pompe's Disease

Exclusion Criteria:

* Those who do not meet inclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subject with Infantile Pompe's Disease seen at Children's between Jan. and February, 2005.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2005-01; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany J Riehle, MD, Principal Investigator — Centers for Disease Control and Prevention